CLINICAL TRIAL: NCT02895308
Title: Differences in Motivation and Adherence to a Prescribed Assignment After Face-to-face and Online Psychoeducation: an Experimental Study
Brief Title: Motivation and Adherence to Psychotherapy Assignments
Acronym: AIDAII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: AIDA-II
Record Dates: First submitted 2016-08-30; First posted 2016-09-09 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-09

CONDITIONS: Behavioral Problems
Keywords: compliance
MeSH Terms: conditions — Problem Behavior; Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Online (Experimental): The Online psychoeducation is presented on on a webpage.
  Interventions: Behavioral: Online psychoeducation
- Face-to-face (Active Comparator): The face-to-face psychoeducation is provided by psychologist and psychology master students.
  Interventions: Behavioral: Face-to-face psychoeducation

INTERVENTIONS:
Behavioral: Online psychoeducation — The online intervention consists of a psychoeducation component taken from affect focused psychotherapy. In this model, emotions are physiological patterns that are shaped mainly in the context of previous relations. By using the model, patients are helped to better understand their current emotions, behaviors and cognitions. The aim of the intervention used in this study is to provide information about the six basic affects and how they may influence everyday behaviors and well-being in recurring patterns.
  Arms: Online
Behavioral: Face-to-face psychoeducation — The intervention consists of a psychoeducation component taken from affect focused psychotherapy. In this model, emotions are physiological patterns that are shaped mainly in the context of previous relations. By using the model, patients are helped to better understand their current emotions, behaviors and cognitions. The aim of the intervention used in this study is to provide information about the six basic affects and how they may influence everyday behaviors and well-being in recurring patterns.
  Arms: Face-to-face

SUMMARY:
The aims of this study are to experimentally investigate and compare whether motivation variables can predict adherence to a prescribed assignment in face-to-face and online interventions using a psychotherapy analogue model.

A total of 100 participants are included in this study and randomized to either a face-to-face or online intervention. Participants in both groups receive a psychoeducation session and are given an assignment for the subsequent week.

DETAILED DESCRIPTION:
The aims of this study are to investigate (1) participants' different forms of motivations to complete a typical psychotherapy assignment, (2) participants' subsequent adherence to the prescribed assignment and the associations between motivations and adherence and (3) any differences regarding motivations, adherence and their associations between the face-to-face and online conditions.

The hypotheses are that participants in the face-to-face condition will report higher motivation as well as higher adherence to the assignments compared to participants in the online condition, that adherence to the assignment will be positively associated with both autonomous motivation and externally regulated motivation and that adherence to the assignment will be more weakly associated with autonomous motivation in the face-to-face compared to the online condition.

To investigate the association between motivation and adherence to assignments in face-to-face and online settings, this study have a longitudinal randomized design with two conditions. The two conditions are face-to-face psychoeducation with a therapist and online psychoeducation with therapist support. A psychotherapy analogue model with a one-session intervention for a non-clinical population is used. Data is collected at baseline and at seven to nine days follow-up.

ELIGIBILITY:
Inclusion Criteria:

* having at least one problematic behavior one wished to understand or change

Exclusion Criteria:

* being below 18 years of age, having no access to a mobile phone and the Internet, reporting elevated levels of depressive symptoms or currently attending psychotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-01; Primary Completion 2015-11 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Adherence to prescribed behavioral assignment | Within 3 days after intervention end.
  The number of prescribed assignments that each participant have completed.

SECONDARY OUTCOMES:
Situational Motivation Scale | Within 3 days after intervention end.
  The SIMS is a self-report measure developed based on the Self-determination theory to measure motivation in experimental tasks.
VAS-scale regarding motivation | Within 3 days after intervention end.
  A Visual Analogue Scale (VAS) measuring homework motivation (scale: 0-100)

CONTACTS AND LOCATIONS:
Overall Officials: Louise Essen, Professor, Study Director — Uppsala University
Locations (1):
- Uppsala University, Uppsala, Uppsala County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alfonsson S, Johansson K, Uddling J, Hursti T. Differences in motivation and adherence to a prescribed assignment after face-to-face and online psychoeducation: an experimental study. BMC Psychol. 2017 Jan 26;5(1):3. doi: 10.1186/s40359-017-0172-5. PMID 28126022